CLINICAL TRIAL: NCT03840967
Title: A Phase II Study Evaluating Safety and Efficacy of Niraparib in Patients With Previously Treated Homologous Recombination (HR) Defective or Loss of Heterozygosity (LOH) High Metastatic Esophageal/Gastroesophageal Junction/Proximal Gastric Adenocarcinoma
Brief Title: A Study Evaluating Safety and Efficacy of Niraparib in Patients With Previously Treated Metastatic Esophageal/Gastroesophageal Junction/Proximal Gastric Adenocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accruals
Sponsor: Shadia Jalal, MD (Other)
Collaborators: GlaxoSmithKline (Industry); Indiana University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Shadia Jalal, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN ESO17-325
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Esophageal Cancer; Gastric Cancer; Adenocarcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Niraparib (Other)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — Niraparib will be administered as a flat-fixed daily dose depending on weight and platelet count. Subjects will take orally on a daily basis for 28 days. Each cycle = 28 days
  Other Names: Zejula

SUMMARY:
Patients can be prescreened for the study at the time of diagnosis of locally advanced or metastatic disease by determining presence of LOH high status and/or deleterious alterations in HR pathway genes in the most recent available tumor tissue sample or in blood if they are found to have germline mutations. Patients with either somatic or germline mutations will be allowed. At the time of disease progression, patients with high LOH or deleterious alterations in HR pathway genes and satisfying all other inclusion criteria will be enrolled on the study. Patients will be treated with niraparib (flat dose) orally every day for 28 days until disease progression, unacceptable side effects, withdrawal of consent, or death. CT of the chest/abdomen/pelvis will be performed every 2 months and response will be assessed by RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. ECOG Performance Status of 0-1 within 14 days prior to registration.
4. Locally advanced esophageal adenocarcinoma or proximal gastric adenocarcinoma or metastatic adenocarcinoma originating from esophagus, GE junction, or proximal stomach who progress/recur beyond 2 months of receiving a platinum- containing regimen

   NOTE: Patients can be pre-screened for study at any time including after surgical resection for locally advanced esophageal cancer, at presentation with metastatic disease and potentially during chemotherapy and radiation prior to surgery.
5. A subject with symptomatic brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic. Patients with asymptomatic brain mets that are untreated will be allowed.
6. Must not have received more than 1 prior line of chemotherapy in the metastatic setting (could have received immunotherapy, VEGF directed therapy, and/or trastuzumab which does not count as chemotherapy).
7. One of the following genetic results is required for eligibility:

   * High LOH in tissue OR
   * HR mutation in tissue OR
   * Germline mutation (blood)

   NOTE: Mutations, deletions or loss by fusions are the acceptable alterations in HR genes as long as they are deleterious. Patients are eligible if they have a mutation in pre-specified HR genes BRCA1/2, PALB2, ATM, BARD1, BRIP1, CDK12, CHEK2, FANCA, RAD51, RAD51B, RAD51C, RAD51D, RAD54L, NBN, ARID1A and GEN1. Deleterious mutations in HR genes are defined as those that have been previously characterized to be loss-of-function/pathogenic/or likely pathogenic as specified per the following databases: Clinvar, OncoKB, or BRCAExchange. Mutations or small insertions or deletions that results in truncation, frameshift, stop codon loss, or stop codon gain will also be considered deleterious irrespective of their presence in the aforementioned databases unless previously characterized to be benign. Copy number losses or disruption by fusion will also be considered deleterious irrespective of their presence in the aforementioned databases. Gene amplifications or variants of unknown significance will not be eligible for inclusion.

   NOTE: Genetic testing results from a CLIA certified lab that confirm one of the following: high LOH in tissue, HR mutation in tissue or germline mutation in blood are required and can be used to meet eligibility. Even if subject has met eligibility with one of the criteria above, results from the other analysis is required if available.

   If prior genetic results are not available, subject must have archival tissue or fresh tissue (by new biopsy) for testing. Both primary tumor tissue and metastatic site sample biopsies are allowed. Blood will also be required for germline mutation analyses. Central confirmation of all results will be performed but are not mandated for eligibility. If a subject has met eligibility with prior genetic results but does not have sufficient archival tissue for central confirmation, a biopsy is not required.
8. Presence of measurable disease by RECIST v1.1, defined as:

   * Tumor lesions that must be accurately measured in at least one dimension (longest diameter in the plane of measurement is to be recorded) with a minimum size of:

     * 10 mm by CT scan (CT scan slice thickness no greater than 5 mm)
     * 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable)
     * 20 mm by chest X-ray
   * Malignant lymph nodes: To be considered pathologically enlarged and measurable, a lymph node must be ≥ 15 mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm). At baseline and in follow-up, only the short axis will be measured and followed.
9. Prior cancer treatment must be completed at least 14 days prior to registration and the subject must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or baseline.
10. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 14 days prior to registration.

    * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
    * Hemoglobin (Hgb) ≥ 9 g/dL
    * Platelet Count (Plt) ≥ 100 K/ mm3
    * Creatinine ≤ 1.5 X upper limit of normal (ULN)
    * Bilirubin ≤ 1.5× ULN ((≤2.0 in patients with known Gilberts syndrome))
    * Aspartate aminotransferase (AST) ≤ 2.5× ULN*
    * Alanine aminotransferase (ALT) ≤ 2.5 × ULN*
11. Females of childbearing potential must have a negative pregnancy test within 7 days prior to study treatment. Urine or serum βhCG if clinically appropriate. If a urine test is done and it is positive or cannot be confirmed as negative, a serum pregnancy test will be required. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
12. Females of childbearing potential must be willing to abstain from heterosexual intercourse or use adequate contraception as described in the protocol. Males must be willing to abstain from heterosexual intercourse or use adequate contraception as described in the protocol.
13. Participants must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.
14. As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.
15. Participant must agree to not donate blood during the study or for 90 days after the last dose of study treatment.

Exclusion Criteria:

1. Prior therapy with a PARP inhibitor
2. Disease progression during first 2 months of standard dose platinum-based chemotherapy (platinum refractory). This excludes low dose platinum based therapy that is given in a chemotherapy-radiation regimen for locally advanced esophageal cancer.
3. Participant must not be simultaneously enrolled in any other interventional clinical trial.
4. Participant must not have had major surgery ≤ 3 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects.
5. Participant must not have received investigational therapy ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy.
6. Participant has had radiation therapy encompassing >20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy.
7. Participant must not have a known hypersensitivity to niraparib components or excipients including tartrazine.
8. Participant must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks prior to initiating protocol therapy.
9. Participant must not have received colony stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony stimulating factor, or recombinant erythropoietin) within 4 weeks prior initiating protocol therapy.
10. Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
11. Participant must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
12. Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.
13. No active secondary cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Michigan Health System, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Niraparib
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Niraparib
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 59 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    ECOG = 0 | 3
    ECOG = 1 | 11
Smoking Status [Count of Participants; unit: Participants]
  Never | 5
  Former | 7
  Current | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the percentage of patients who reached CR or PR by RECIST 1.1.
Time Frame: Up to maximum of 5 months.
Population: Out of 14 patients, three patients were not evaluable for best response.
Measure: Number; unit: Percentage of participants
Arm/Group | Niraparib
Number analyzed (Participants) | 11
Percentage of participants | 0

2. Secondary Outcome: Adverse Events
Description: Number of participants with treatment related adverse events are reported by CTCAEv5 term and grade.
Time Frame: AE had been recorded from time of signed informed consent until 30 days after discontinuation of study drug(s) or until a new anti-cancer treatment starts, whichever occurs first, up to a maximum of 6 months.
Measure: Number; unit: Participants
Arm/Group | Niraparib
Number analyzed (Participants) | 14
Participants
  Anemia | 7
  Fatigue | 7
  Platelet count decreased | 7
  Nausea | 6
  Headache | 5
  White blood cell decreased | 5
  Anorexia | 3
  Constipation | 3
  Weight loss | 3
  Abdominal pain | 2
  Diarrhea | 2
  Dizziness | 2
  Dyspepsia | 2
  Hypocalcemia | 2
  Lymphocyte count decreased | 2
  Neutrophil count decreased | 2
  Vomiting | 2
  Arthralgia | 1
  Aspartate aminotransferase increased | 1
  Cough | 1
  Dry mouth | 1
  Dry skin | 1
  Dysgeusia | 1
  Dyspnea | 1
  Hypercalcemia | 1
  Hyponatremia | 1
  Sinus tachycardia | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time from treatment start until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Up to a maximum of 5 months.
Population: Out of 14 patients, three patients were not evaluable for PFS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Niraparib
Number analyzed (Participants) | 11
Months | 1.8 [1 to 3.7]

4. Secondary Outcome: Disease Control Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Disease control rate (DCR) is defined as the percentage of evaluable patients with stable disease (SD) for 8 weeks, or partial response (PR), or complete response (CR) according to RECIST 1.1.
Time Frame: Up to maximum of 5 months.
Population: Out of 14 patients, three patients were not evaluable for DCR.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Niraparib
Number analyzed (Participants) | 11
Percentage of participants | 18.2 [2.3 to 51.8]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 24 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 6 months.
Arm/Group | Niraparib
All-Cause Mortality (participants affected / at risk) | 12/14
Serious Adverse Events (participants affected / at risk) | 3/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib (N=14)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Niraparib (N=14)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (5)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 5 (7)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 10 (23)
ANOREXIA (Metabolism and nutrition disorders) | 4 (8)
ANXIETY (Psychiatric disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (5)
CHILLS (General disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 6 (6)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
CREATININE INCREASED (Investigations) | 3 (4)
DIARRHEA (Gastrointestinal disorders) | 3 (5)
DIZZINESS (Nervous system disorders) | 3 (4)
DRY MOUTH (Gastrointestinal disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 3 (4)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
EOSINOPHILIA (Blood and lymphatic system disorders) | 1 (1)
FATIGUE (General disorders) | 10 (13)
FEVER (General disorders) | 3 (6)
HEADACHE (Nervous system disorders) | 8 (11)
HEPATIC INFECTION (Infections and infestations) | 1 (2)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (3)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (6)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (Infections and infestations) | 1 (2)
INSOMNIA (Psychiatric disorders) | 3 (3)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 2 (7)
LUNG INFECTION (Infections and infestations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (2)
MEMORY IMPAIRMENT (Nervous system disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (3)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 7 (14)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (6)
PAIN (General disorders) | 2 (3)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 8 (11)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (1)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (3)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SURGICAL AND MEDICAL PROCEDURES - OTHER, SPECIFY (Surgical and medical procedures) | 4 (6)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
VOMITING (Gastrointestinal disorders) | 3 (5)
WEIGHT LOSS (Investigations) | 4 (4)
WHITE BLOOD CELL DECREASED (Investigations) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT03840967/Prot_SAP_000.pdf